CLINICAL TRIAL: NCT05563064
Title: Effect of Herbal Formulation on Karika Syrup on Thrombocytes Count
Brief Title: Effect of Herbal Formulation on Thrombocytes Count
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shifa Ul Mulk Memorial Hospital (Other)
Responsible Party: Principal Investigator, Dr. Hafiz Muhammad Asif, Chairperson Department of Eastern Medicine, Jinnah University, Shifa Ul Mulk Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Shayan Fatima
Record Dates: First submitted 2022-09-28; First posted 2022-10-03 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Thrombocytopenia
Keywords: Thrombocyte Count, Karika
MeSH Terms: conditions — Thrombocytopenia

STUDY DESIGN:
Intervention Model Description: A randomized, open, prospective, multicenter clinical trial to evaluate the effects of Karika syrup on complete blood count specifically thrombocytes (platelets)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Karika Syrup (Experimental): Karika syrup has been used to treat thrombocytopenia
  Interventions: Drug: Karika Syrup

INTERVENTIONS:
Drug: Karika Syrup — To evaluate the effects of Karika syrup on complete blood count specifically thrombocytes (platelets) collected from blood samples of patients after treatment of 15 days long period.

SUMMARY:
Effect of Herbal Formulation Karika Syrup on Thrombocyte Count.

DETAILED DESCRIPTION:
In this study, we will evaluate the effect of Herbal Formulation Karika (composed of Carica papaya leaf extract and Tinosporacordifolia) on Complete Blood Count, specifically on Platelet Count. Low Platelet Count is highly observant during multiple diseases namely dengue, malaria, typhoid, chikungunya, viral infections, and other Diseases.

The proposed study is a randomized, open, prospective, multicenter clinical trial. Extracts found in Karika syrup are beneficial in escalating platelet count, and also have anti-inflammatory and antipyretic activity. The therapeutic indication of Karika is proven through this clinical study in patients with low platelet count associated with dengue, typhoid, malaria, viral fever, and chikungunya fever.

Dengue is a tropical disease caused by the RNA virus which resides in mosquitoes. Symptoms include high-grade fever, visual disturbances, pain in the eyes and head, nausea, vomiting, musculoskeletal pain, stiffness of joints, mild to moderate and severe bleeding, and sometimes puerperal rash appearing on the skin due to a deficiency of thrombocytes.

The Chikungunya virus is spread by the bite of an infected mosquito. Typhoid is caused by Salmonella typhi a bacterium. Typhoid fever symptoms are seen widely in the human body that may observe from relatively minor cases of diarrhea with low-grade fever to high-grade fever and profound diarrhea with involvement of multiple systems.1

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

  1. Female and Male patients of age 14 to 60 years.
  2. Patient suffering from complaints of Weakness, Fatigue, Puerperal Rashes, Shortness of Breath, Low Hemoglobin, and History of Fever on & off, Epistaxis.18
  3. Patients from Karachi and Kapri Mori(Labors, Employed, Multigravida females, Housewives, Domestic helpers, Working women, School, College, and University Students).
  4. All socioeconomic classes are included in the study.
  5. Patients having a history of Covid-19, Viral fever, Typhoid, and other illnesses in which there has been a low platelet count.2

Exclusion Criteria:

* Exclusion Criteria:

  1. Pregnant females are excluded.17
  2. Patients with co-morbidities like uncontrolled hypertension and liver disorder are excluded.4,5,6
  3. Patient having known drug reaction from any content of formulation is excluded.7
  4. Patients suffering from serious illnesses like encephalitis, coma, meningitis, or head injury that make them bedridden or hospitalized are excluded.4,6

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
EFFECT OF HERBAL FORMULATION KARIKA SYRUP ON THROMBOCYTE COUNT | 3 years
  This study is designed to check or confirm the Karika syrup efficacy for increasing the platelet count, its anti-inflammatory and anti-pyretic actions. This medicinal use of Karika will be confirmed through clinical studies in patients with low platelet count associated with dengue, typhoid, malaria, viral fever& chikungunya fever.9 It is based on the interpretations as generated from CBC by analyzing it on SPSS. 10 It is research-based open, randomized clinical trial on 72 subjects Multi-centered: Karachi (Kalaboard, Jafar-e-tyyar) and Interior Sindh (Kapri Mori).

CONTACTS AND LOCATIONS:
Locations (1):
- Pakistan, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided